CLINICAL TRIAL: NCT05009446
Title: A Prospective Single Arm Clinical Study of Induction Chemoradiotherapy Combined With Surgery in the Treatment of Locally Advanced Sinonasal Malignant Melanoma
Brief Title: Single Arm Study of Induction Chemoradiotherapy Combined With Surgery in the Treatment of Locally Advanced SNMM
Acronym: SNMM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hongmeng Yu, Principal Investigator,Head of Rhinology, Eye & ENT Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNMM-SA-RTNeo
Record Dates: First submitted 2021-07-18; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Mucosal Melanoma; Sinonasal Melanoma
Keywords: Sinonasal mucosal melanoma; Inductive radiotherapy; chemotherapy; overall survival
MeSH Terms: interventions — Endoscopy; Radiotherapy, Intensity-Modulated; Protons; Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative radiotherapy and chemotherapy (Experimental): Preoperative radiotherapy and chemotherapy plus endoscopic surgery
  Interventions: Procedure: endoscopic surgery; Radiation: intensity-modulated radiation therapy or volume of rotating intensity-modulated radiotherapy or Proton or heavy ion radiation therapy; Drug: Chemotherapy drug

INTERVENTIONS:
Procedure: endoscopic surgery — endoscopic surgery or endoscope-assisted surgery open surgery
Radiation: intensity-modulated radiation therapy or volume of rotating intensity-modulated radiotherapy or Proton or heavy ion radiation therapy — radiotherapy was administrated before surgery
Drug: Chemotherapy drug — Chemotherapy was administrated before surgery. Chemotherapy may also be administrated after surgery in selected cases.

SUMMARY:
Sinonasal mucosal melanoma (SNMM) is a very rare tumor, and SNMM is highly aggressive in nature, with a 5-year survival rate of about 20~30%. Most patients underwent local recurrence and distant metastasis within one or two years of treatment.

There is no unified standard for the treatment of SNMM.The principle of treatment for surgically resectable stage T3 and partial T4 SNMM is complete resection of the primary tumor, combined with postoperative radiotherapy. While locally unresectable SNMM has a poorer prognosis, lower incidence, fewer clinical data have been reported.

This study will explore the role of preoperative radiotherapy and chemotherapy in improving the 2-year OS rate, loco-regional control rate and distant metastasis rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old;
2. Pathologically confirmed with sinonasal mucosal melanoma;
3. Eligible for assessment by enhanced contrast computed tomography scan or magnetic Resonance Imaging (MRI);
4. T4N0-1M0 according to the 8th edition American Joint Committee on Cancer (AJCC) staging system, and breaks through the natural anatomical boundaries of orbital fascia or dura mater; or 2) any Tumor stage, with retropharyngeal node metastasis. unresectable tumor after multi-disciplinary team (MDT) discussion.
5. Eastern Cooperative Oncology Group (ECOG) score between 0 to 2;
6. No distant metastasis;
7. Adequate organ function;
8. Sign the informed consent forms.

Exclusion Criteria:

1. There is evidence or suspicious of distant metastasis on clinical examination or imaging examination;
2. suffered from uncontrolled concurrent diseases that may interfere with treatment;
3. Suffered from another malignant tumor or multiple primary tumors at the same time within 5 years (excluding fully treated basal cell or squamous cell skin cancer, cervical cancer in situ, etc.);
4. With surgical contraindications: severe cardiopulmonary disease, coagulation dysfunction, etc;
5. With and conditions that interfere with patient compliance or safety;
6. With severe mental or neurological diseases;
7. Uncontrolled active infection diseases;
8. Pregnant or breastfeeding women;
9. Patients without personal freedom or independent civil capacity;
10. Other situations that are not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-08-10 (Estimated); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of first treatment until the date of death from any cause,through study completion,up to 2 years.
  2 year Overall Survival rate

SECONDARY OUTCOMES:
Progression-free survival | From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first，through study completion,up to2 years
  the date of first treatment to the first recording of disease progression or death from any cause.
Local progression free survival | From date of first treatment to local failure or date of death from any cause,through study completion,up to 2 years
  the date of first treatment to local failure or death
Regional progression free survival | From date of first treatment to regional failure or date of death from any cause, through study completion,up to 2 years
  the date of first treatment to regional failure or death
Distant metastasis free survival | From date of first treatment to distant metastasis or date of death from any cause, through study completion,up to 2 years
  the date of first treatment to distant metastasis or death
ORR | From date of first treatment to the date of best overall response before surgery, assessed up to 6 months
  objective remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, MD,PhD, Principal Investigator — Eye& ENT Hospital of Fudan University, Shanghai, China
Locations (1):
- Eye& ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China